CLINICAL TRIAL: NCT01738516
Title: Contribution of High Resolution EEG Functional Connectivity Measures to Presurgical Evaluation of Patients With Intractable Epilepsy
Acronym: conneXion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-A01227-36; LOC/12-07 (Other: Rennes University Hospital (Direction of Clinical Research))
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- epileptic patients (Other): Electroencephalography
  Interventions: Procedure: Electroencephalography
- Healthy Volunteers (Other): Electroencephalography and additional experimental tasks
  Interventions: Procedure: Electroencephalography and additional experimental tasks

INTERVENTIONS:
Procedure: Electroencephalography — Epileptic patients, as in healthy volunteers will be offered a review of EEG recording equipment resting on EEG-HR 256-channel EGI © in operation since January 2012 in the Van Gogh Service Unit of Neurology Rennes University Hospital (hospital Pontchaillou). The EEG is a routine now included in the Phase I report some epileptic patients during presurgical investigation. Patients to be included in this research protocol pass all review on the new device EEG-HR 256 channels. In addition to the rest condition, shared by both groups of participants, the healthy control subjects participate in two additional experimental tasks to be performed during recording. A picture naming task and a task of spelling words represented by these images.
  Arms: epileptic patients
Procedure: Electroencephalography and additional experimental tasks — Epileptic patients, as in healthy volunteers will be offered a review of EEG recording equipment resting on EEG-HR 256-channel EGI © in operation since January 2012 in the Van Gogh Service Unit of Neurology Rennes University Hospital (hospital Pontchaillou). The EEG is a routine now included in the Phase I report some epileptic patients during presurgical investigation. Patients to be included in this research protocol pass all review on the new device EEG-HR 256 channels. In addition to the rest condition, shared by both groups of participants, the healthy control subjects participate in two additional experimental tasks to be performed during recording. A picture naming task and a task of spelling words represented by these images.
  Arms: Healthy Volunteers

SUMMARY:
Electroencephalography (EEG) with very high spatial resolution (HR-EEG, 256 electrodes) allow for better analysis of local and global activity of the cerebral cortex, as compared with conventional EEG. Since January 2012, the Neurology Department of CHU Rennes is the first clinical service in France equipped with such a system.

Applied to HR-EEG recordings, brain connectivity methods are likely to provide essential information (in the form of "connectivity graphs") on cortical networks, either dysfunctional or not, involved in the generation of interictal paroxysms (like spikes or spike-waves) and during seizures.

So far, many methods have been proposed (see for a review: Wendling et al., 2009; Wendling et al., 2010). However, since each method is highly sensitive to the type of model that is assumed for the underlying relationship between distinct brain regions (Ansari-Asl et al., 2006), none of them has yet demonstrated its effectiveness.

ELIGIBILITY:
Inclusion Criteria Patients:

* Being more than 18 years old,
* Having a chronic partial epilepsy resistant to medical treatments well administered and well followed in the course of pre-surgical assessment.

Inclusion Criteria Healthy Volunteers:

* Being French native speaker,
* Being more than 18 years old,
* Being right-handed.

Exclusion Criteria Patients:

* All patients for whom a preoperative surgical exam is not suitable,
* Any patient with psychiatric disease or intellectual disorder such that informed consent could not be obtained,
* Any patient with no abnormal EEG during intercritical phases,
* All patients presenting psychiatric, neuropsychological or developmental difficulties in addition to epilepsy,
* Adult persons subject to legal protection (judicial protection, temporary guardianship/guardianship, administrative supervision), persons deprived of their liberty and pregnant or lactating women.

Exclusion Criteria Healthy Volunteers:

* The presence of any psychiatric, neuropsychological, and developmental disorder,
* Any uncorrected visual impairment,
* Any trouble or delay in learning to read / speak or write French,
* Being fully bilingual or multilingual
* Medication, treatment and / or substances that may alter or modify brain functions,
* Adult persons subject to legal protection (judicial protection, temporary guardianship/guardianship, administrative supervision), persons deprived of their liberty and pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The quality of matching between i) the graphs produced by the evaluated connectivity method(s) applied to the HR-EEG and ii) the results of the visual analysis typically performed by an expert on the standard EEG recorded during intercritical phase. | 2 years
  Main objective :To determine which functional connectivity estimation method(s) show(s) best performance(s) for the identification of epileptogenic networks from the HR-EEG recording performed in epileptic patients.

SECONDARY OUTCOMES:
The quality of matching between i) the connectivity graphs obtained from control subjects performing a well defined cognitive task to ii) data from the literature on networks activated and sustaining these cognitive processes. | 2 years
  Our secondary objectives are:
  * The application of linear, non-linear and phase synchronization methods in digital signal processing on broadband band analysis or on band-filtered EEG signals acquired during HR-EEG explorations of patients with epilepsy,
  * The evaluation of the performance of these methods by comparing the resulting connectivity graphs with those expected in healthy subjects (controls),
  * The application of the methods offering the best performances to data acquired in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Biraben, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France

REFERENCES:
- [Result] Mheich A, Hassan M, Khalil M, Gripon V, Dufor O, Wendling F. SimiNet: A Novel Method for Quantifying Brain Network Similarity. IEEE Trans Pattern Anal Mach Intell. 2018 Sep;40(9):2238-2249. doi: 10.1109/TPAMI.2017.2750160. Epub 2017 Sep 8. PMID 28910755
- [Result] Kabbara A, El Falou W, Khalil M, Wendling F, Hassan M. The dynamic functional core network of the human brain at rest. Sci Rep. 2017 Jun 7;7(1):2936. doi: 10.1038/s41598-017-03420-6. PMID 28592794
- [Result] Mheich A, Hassan M, Khalil M, Berrou C, Wendling F. A new algorithm for spatiotemporal analysis of brain functional connectivity. J Neurosci Methods. 2015 Mar 15;242:77-81. doi: 10.1016/j.jneumeth.2015.01.002. Epub 2015 Jan 10. PMID 25583381
- [Result] Hassan M, Merlet I, Mheich A, Kabbara A, Biraben A, Nica A, Wendling F. Identification of Interictal Epileptic Networks from Dense-EEG. Brain Topogr. 2017 Jan;30(1):60-76. doi: 10.1007/s10548-016-0517-z. Epub 2016 Aug 22. PMID 27549639
- [Result] Rizkallah J, Benquet P, Kabbara A, Dufor O, Wendling F, Hassan M. Dynamic reshaping of functional brain networks during visual object recognition. J Neural Eng. 2018 Oct;15(5):056022. doi: 10.1088/1741-2552/aad7b1. Epub 2018 Aug 2. PMID 30070974
- [Result] Hassan M, Shamas M, Khalil M, El Falou W, Wendling F. EEGNET: An Open Source Tool for Analyzing and Visualizing M/EEG Connectome. PLoS One. 2015 Sep 17;10(9):e0138297. doi: 10.1371/journal.pone.0138297. eCollection 2015. PMID 26379232
- [Result] Hassan M, Dufor O, Merlet I, Berrou C, Wendling F. EEG source connectivity analysis: from dense array recordings to brain networks. PLoS One. 2014 Aug 12;9(8):e105041. doi: 10.1371/journal.pone.0105041. eCollection 2014. PMID 25115932
- [Result] Hassan M, Benquet P, Biraben A, Berrou C, Dufor O, Wendling F. Dynamic reorganization of functional brain networks during picture naming. Cortex. 2015 Dec;73:276-88. doi: 10.1016/j.cortex.2015.08.019. Epub 2015 Sep 28. PMID 26478964